CLINICAL TRIAL: NCT04293627
Title: ADAPTING AND IMPLEMENTING AN INTEGRATED CARE MODEL FOR YOUTH WITH AUTISM SPECTRUM DISORDER AND PSYCHIATRIC COMORBIDITY
Brief Title: Access to Tailored Autism Integrated Care Pilot Study
Acronym: ATTAIN
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: Kaiser Permanente (Other); San Ysidro Health Center (Other); Rady Children's Hospital, San Diego (Other)
Responsible Party: Principal Investigator, Nicole Stadnick, Assistant Professor, University of California, San Diego
Other Study IDs: UC San Diego
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Autism Spectrum Disorder; Mental Health Issue
Keywords: pediatric primary care; implementation science; co-occurring mental health conditions; community academic partnership
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: ATTAIN — ATTAIN is an 8-step model to identify co-occurring mental health conditions and facilitate linkage to mental health services for youth with an existing autism spectrum disorder diagnosis.

SUMMARY:
Children with autism spectrum disorder (ASD) represent a rapidly growing, high-priority clinical population highlighted by the NIMH and Interagency Autism Coordinating Committee due, in part, because they have multiple service needs including access to effective mental health treatment given high rates of psychiatric comorbidities. Pediatric primary care is a critical and ongoing point of health care access for children with ASD and thus represents an ideal setting for identification of mental health service needs and appropriate linkage to care. The proposed study will use implementation science theory and methods and a research-community partnership approach to: 1) identify targets to improve mental health screening and linkage to mental health services in primary care for children with ASD, 2) adapt integrated care procedures into "Access To Tailored Autism INtegrated Care," ATTAIN, to facilitate identification of mental health problems and linkage to evidence-based care for youth with ASD, and 3) conduct an open trial feasibility pilot test of ATTAIN in pediatric primary care.

DETAILED DESCRIPTION:
This description is focused solely on the feasibility pilot test of ATTAIN in pediatric primary care.

Phase 3. Conduct an open trial feasibility pilot test of ATTAIN (directly informed by adaptations identified earlier in the larger study) in pediatric primary care.

Participants

Providers: A total of 45 pediatric care providers and staff will be recruited for enrollment from primary care practices in the region. This targeted sample size was chosen based on sample sizes used within completed pilot studies focused on service interventions in pediatric care. Each provider and healthcare staff member will be asked to use or support use of ATTAIN with up to 5 eligible patients over four months.

Families: Eligible pediatric patients must be: 1) English and/or Spanish-speaking, 2) between 4-16 years of age and 3) have a documented ASD diagnosis in the electronic health record. After four months of ATTAIN use by their child's primary care provider, caregivers will be contacted by the research team to be invited to complete an online survey about their child's healthcare experiences over the past four months.

Procedure Leadership at each primary care organization will be approached about their primary care practices participating in the pilot study. Primary care practices within each organization will be purposively selected for targeted recruitment of providers for ATTAIN implementation based on volume of patients with ASD. Members of the research team will request an invitation to present at regularly scheduled staff meetings to recruit primary care providers. Interested providers will be asked to complete a study interest form and indicate preferred times to attend a group meeting to review study participation details, the Study Information Sheet, and receive training in using the ATTAIN model. For some clinics, leadership may prefer that the recruitment and training be conducted during the same meeting for the purpose of reducing staff burden. At these meetings, the research team will provide a meal and refreshments. Subsequently, trained providers will be asked to use ATTAIN with up to 5 eligible patients during any outpatient appointment (e.g., annual check-ups, drop-in appointments) to maximize early detection of mental health problems and opportunity to link to mental health services. Throughout the 4 months, we may ask providers and supporting staff to elaborate on their experiences using ATTAIN via e-mail or phone-call to understand challenges to implementation, recommendations for improving implementation or adaptations in implementing the ATTAIN model in their clinic. Time to complete these brief reflections will take no more than 5-10 minutes each. Quantitative data of ATTAIN use will be extracted from patient charts and de-identified data will be sent to the research team during the four month study period and at the end of 4 months. After 4 months of ATTAIN delivery, participating providers and caregivers of youth with ASD with whom providers used ATTAIN will be asked to complete a brief online survey regarding their experiences using ATTAIN. Providers and staff will be asked to attend a meeting, where food and light refreshments will be provided, to complete the survey. In addition, providers and staff will be invited to participate in a post-study interview that will be offered to be completed by phone or in-person. Caregivers will receive $20 for survey completion. The ATTAIN model was developed to be embedded within routine primary care settings and workflow so there are minimal risks to primary care providers, caregivers or children associated with participation.

ELIGIBILITY:
Providers: A total of 45 pediatric care providers and staff will be recruited for enrollment from primary care practices in the region. This targeted sample size was chosen based on sample sizes used within completed pilot studies focused on service interventions in pediatric care. Each provider and healthcare staff member will be asked to use or support use of ATTAIN with up to 5 eligible patients over four months.

Families: Eligible pediatric patients must be: 1) English and/or Spanish-speaking, 2) between 4-16 years of age and 3) have a documented ASD diagnosis in the electronic health record. After four months of ATTAIN use by their child's primary care provider, caregivers will be contacted by the research team to be invited to complete an online survey about their child's healthcare experiences over the past four months.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Providers and families will be recruited from pre-identified pediatric primary care clinics in Southern California serving children with autism spectrum disorder.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability of ATTAIN | Post-pilot (4 months of ATTAIN delivery)
  The Perceived Characteristics of Intervention Scale (PCIS) will be used to examine providers' and staff's perspectives regarding feasibility and acceptability of ATTAIN. The PCIS is a 20-item scale that assesses attitudes towards a specific intervention including relative advantage, compatibility, and complexity. Participants are asked to rate the extent to which they agree with each item on a 5-point Likert scale. Example items include, "The ATTAIN model is clear and understandable" and "Using the ATTAIN model fits well with the way I like to work."
Acceptability of Intervention Measure | Post-pilot (4 months of ATTAIN delivery)
  A 4-item measure to assess the extent to which providers/staff believe ATTAIN is acceptable.
Feasibility of Intervention Measure | Post-pilot (4 months of ATTAIN delivery)
  A 4-item measure to assess the extent to which providers/staff believe ATTAIN is feasible.
ASD + Mental Health Comfort and Knowledge Questionnaire | Post-pilot (4 months of ATTAIN delivery)
  A questionnaire adapted from autism implementation studies (Brookman-Frazee et al., 2019; Stadnick et al., 2020) assessing provider perceptions of comfort and knowledge about serving children with ASD.
Measure of Innovation-Specific Implementation Intentions (MISII) | Post-pilot (4 months of ATTAIN delivery)
  A 3-item measure assessing provider intentions to use a specific innovation (ATTAIN).

SECONDARY OUTCOMES:
ATTAIN Uptake | Post-pilot (4 months of ATTAIN delivery)
  ATTAIN uptake will be measured using extracted data from the electronic health record system or provider-reported data about the number of patients with whom they used ATTAIN. Specifically, uptake will be defined as the proportion of ATTAIN-eligible patients (i.e., children with a documented ASD diagnosis) to the number children with whom providers used ATTAIN.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole A Stadnick, PhD, MPH, Principal Investigator — Assistant Professor
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
Researchers may contact the PI to request de-identified data in aggregate form, as appropriate.

REFERENCES:
- [Background] Stadnick NA, Brookman-Frazee L, Mandell DS, Kuelbs CL, Coleman KJ, Sahms T, Aarons GA. A mixed methods study to adapt and implement integrated mental healthcare for children with autism spectrum disorder. Pilot Feasibility Stud. 2019 Mar 28;5:51. doi: 10.1186/s40814-019-0434-5. eCollection 2019. PMID 30976456
- [Background] Broder-Fingert S, Stadnick NA, Hickey E, Goupil J, Diaz Lindhart Y, Feinberg E. Defining the core components of Family Navigation for autism spectrum disorder. Autism. 2020 Feb;24(2):526-530. doi: 10.1177/1362361319864079. Epub 2019 Jul 16. PMID 31311287
- [Background] Stadnick NA, Martinez K, Aarons GA, Lee DA, Van Cleave J, Brookman-Frazee L. Pediatric Primary Care Perspectives on Integrated Mental Health Care for Autism. Acad Pediatr. 2020 Nov-Dec;20(8):1140-1147. doi: 10.1016/j.acap.2020.03.006. Epub 2020 Mar 20. PMID 32205263
- [Background] Stadnick NA, Lau AS, Dickson KS, Pesanti K, Innes-Gomberg D, Brookman-Frazee L. Service use by youth with autism within a system-driven implementation of evidence-based practices in children's mental health services. Autism. 2020 Nov;24(8):2094-2103. doi: 10.1177/1362361320934230. Epub 2020 Jul 18. PMID 32686469

DOCUMENTS (1):
  • Informed Consent Form (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT04293627/ICF_000.pdf